CLINICAL TRIAL: NCT01930110
Title: An Open-label, Randomized, Cross-over Study to Compare the Efficacy of Single-hormone Closed-loop Strategy and Dual-hormone Closed-loop Strategy at Regulating Glucose Levels During Continuous Exercise and Interval Exercise in Adults With Type-1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) During Exercise in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Société Francophone du Diabète (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-06
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Insulin; Glucagon; Closed-loop system; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-hormone closed-loop system (Active Comparator): In single-hormone closed-loop system, variable subcutaneous insulin infusion rate will be used to regulate glucose levels
  Interventions: Other: 60-minute exercise; Other: 40-minute interval exercise
- Dual-hormone closed-loop system (Active Comparator): In dual-hormone closed-loop system, variable subcutaneous insulin and glucagon infusion rates will be used to regulate glucose levels
  Interventions: Other: 60-minute exercise; Other: 40-minute interval exercise

INTERVENTIONS:
Other: 60-minute exercise — Patients will be admitted at the research clinical facility at 14:30. Closed-loop strategy will start at 15:30. At 18:00, patients will performed a 60-minute exercise at 60% of VO2 max. Patients will be discharged at 20:00.
Other: 40-minute interval exercise — Patients will be admitted at the research clinical facility at 14:30. Closed-loop strategy will start at 15:30. At 18:00, patients will performed a 40-minute interval exercise. Patients will be discharged at 20:00.

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

The objective is to compare the efficacy of single-hormone closed-loop strategy and dual-hormone closed-loop strategy at regulating glucose levels during continuous exercise and interval exercise.

The investigator hypothesized that dual-hormone closed-loop strategy is superior to single-hormone closed-loop strategy in regulating glucose levels during exercise periods.

DETAILED DESCRIPTION:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

We aim to conduct a randomized two-way cross-over trial comparing single-hormone closed-loop strategy and dual-hormone closed-loop strategy to compare the two interventions during exercise periods in adults with type 1 diabetes. A moderate intensity exercise will be performed for 60 minutes at 60% of the maximum oxygen consumption (VO2max). A high intensity exercise will be 40 minutes of interval training. The interval training will be preceded by a 10 minutes warm-up and followed by a 10 minutes cool down.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of old.
* Clinical diagnosis of type 1 diabetes for at least one year.
* The subject will have been on insulin pump therapy for at least 3 months.
* Last (less than 3 months) HbA1c ≤ 12%.

Exclusion Criteria:

* Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
* Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* Ongoing pregnancy.
* Severe hypoglycemic episode within two weeks of screening.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
* Failure to comply with team's recommendations (e.g. not willing to eat snack, not willing to change pump parameters, etc).
* Problems with venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The number of patients experiencing exercise-induced hypoglycemia requiring dextrose infusion (< 3.3 mmol/L symptomatic or < 3.0 mmol/L regardless of symptoms). | 18:00 hours to 19:30 hours

SECONDARY OUTCOMES:
Decrease in glucose levels during each exercise | 18:00 to 19:30 hours or 18:00 to 19:10 depending on the exercise performed
  Difference between glucose levels at the beginning of the exercise and the lowest glucose level from the start of the exercise until 30 minutes after exercise).
Area under the curve of plasma glucose levels < 4 mmol/L | 15:30 hours to 19:30 hours
Percentage of time of plasma glucose levels < 4 mmol/L | 15:30 hours to 19:30 hours
Number of patients with an exercise-induced hypoglycemia < 3.9 mmol/L | 15:30 hours to 19:30 hours
Decremental area under the curve from the start of the exercise for 90 minutes. | 18:00 to 19:30
Percentage of time-in-target defined as between 4 and 10 mmol/L | 15:30 hours to 19:30 hours
Mean time (minutes) to the first hypoglycemic event during the exercise period | 18:00 to 19:00
The amount of dextrose infused | 15:30 to 19:30

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Taleb N, Emami A, Suppere C, Messier V, Legault L, Ladouceur M, Chiasson JL, Haidar A, Rabasa-Lhoret R. Efficacy of single-hormone and dual-hormone artificial pancreas during continuous and interval exercise in adult patients with type 1 diabetes: randomised controlled crossover trial. Diabetologia. 2016 Dec;59(12):2561-2571. doi: 10.1007/s00125-016-4107-0. Epub 2016 Oct 4. PMID 27704167